CLINICAL TRIAL: NCT02152384
Title: The Effect of Treatment With Basal Insulin Peglispro or Insulin Glargine on the Dose Response Effect of Prandial Insulin Lispro in Patients With Type 1 Diabetes Mellitus.
Brief Title: A Study to Compare and Measure the Effects of Insulin Peglispro (LY2605541) and Glargine on Meal Time Insulin Requirements
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15406; I2R-MC-BIDU (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-05-28; First posted 2014-06-02 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — basal insulin peglispro; LY2605541; Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin peglispro (LY2605541, with Insulin Lispro) (Experimental): Insulin peglispro (LY2605541) once daily subcutaneous (SC) injection at bedtime. Insulin lispro given SC prandially or as bolus as required
  Interventions: Drug: Insulin Peglispro; Drug: Insulin Lispro
- Insulin Glargine (with Insulin Lispro) (Active Comparator): Insulin glargine once daily SC injection at bedtime. Insulin lispro given SC prandially or as a bolus as required
  Interventions: Drug: Insulin Lispro; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Peglispro — Administered SC
  Other Names: LY2605541
  Arms: Insulin peglispro (LY2605541, with Insulin Lispro)
Drug: Insulin Lispro — Administered SC
Drug: Insulin Glargine — Administered SC
  Arms: Insulin Glargine (with Insulin Lispro)

SUMMARY:
This study will look into how a base dose of insulin peglispro and insulin glargine will affect the meal time dose and efficacy of insulin lispro in type 1 diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Have a stable (within 0.5 percent (%) from last measure) glycated hemoglobin (HbA1c) <9.0%
* Have a stable (within 30%) basal insulin dose of 0.2 to 1.0 units per kilogram per day (U/kg/day) and a total daily insulin dose (basal + prandial/bolus) <1.5 units per kilogram (U/kg)
* Have C-peptide <0.3 nanomoles per liter (nmol/L)
* Are able and willing to eat the protocol specified standard breakfast and other meals as required

Exclusion Criteria:

* Have corrected QT interval (QTc) prolongation >500 milliseconds (ms) or have any other abnormality in the 12 lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure as determined by the investigator
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (apart from Type 1 Diabetes Mellitus [T1DM]), hematological, or neurological disorders
* Have fasting triglycerides (TGs) >400 milligrams per deciliter (mg/dL) (4.52 micromoles per liter [mmol/L])
* Have used systemic corticosteroids within 4 weeks prior to randomization
* Currently receive insulin pump or insulin degludec
* Have poorly controlled diabetes or are known to have poor awareness of hypoglycemia
* Have history of gastroparesis or gastrointestinal malabsorption
* Require treatment with any drug other than insulin to treat diabetes
* Have a previous history of proliferative retinopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuss, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A/B: Treatment A: Insulin peglispro (LY2605541) once daily subcutaneous (SC). Insulin lispro given SC prandially or as bolus as required
  Treatment B: Insulin glargine once daily subcutaneous (SC). Insulin lispro given SC prandially or as bolus as required
- Treatment Sequence B/A: Treatment B: Insulin glargine once daily subcutaneous (SC). Insulin lispro given SC prandially or as bolus as required
  Treatment A: Insulin peglispro (LY2605541) once daily subcutaneous (SC). Insulin lispro given SC prandially or as bolus as required
Period: Run In (1-5 Week Transition)
Arm/Group | Treatment Sequence A/B | Treatment Sequence B/A
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Period 1
Arm/Group | Treatment Sequence A/B | Treatment Sequence B/A
Started | 14 | 14
Received at Least 1 Dose of Study Drug | 14 | 14
Completed | 13 | 12
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 1
Period: Period 2
Arm/Group | Treatment Sequence A/B | Treatment Sequence B/A
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All randomized participants who received at least 1 dose of study drug.
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 28

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics (PD): Plasma Glucose Area Under the Concentration Curve Zero Through 5 Hours (AUC 0-5h), Above Pre Meal Baseline for Insulin Lispro
Description: To quantitate the pharmacodynamic (PD) effect of a range of prandial insulin lispro doses after treatment with insulin peglispro (LY2605541) compared to insulin glargine during a meal tolerance test (MTT), with sequenced doses of insulin lispro ranging from 25% to 150% of each participant's normal dose. Data presented as hours times milligrams per deciliter (mg*h/dL)
Time Frame: Day 30, 31, 32, 33, 34, pre-breakfast and10,20,30,40,50,60,90,120,150,180,210,240,270, 300 minutes (5 hours) post-breakfast
Population: All participants who received at least 1 dose of study drug and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Groups:
- Insulin Peglispro (LY2605541): Insulin peglispro (LY2605541) administered SC daily
- Insulin Glargine: Insulin glargine administered SC daily
Arm/Group | Insulin Peglispro (LY2605541) | Insulin Glargine
Number analyzed (Participants) | 27 | 26
mg*h/dL
  25% Normal Dose | 677.84 (146.48) | 716.52 (179.89)
  50% Normal Dose: number analyzed (Participants) | 26 | 25
  50% Normal Dose | 572.96 (149.76) | 506.22 (188.54)
  75% Normal Dose: number analyzed (Participants) | 27 | 25
  75% Normal Dose | 393.28 (175.68) | 369.08 (169.08)
  100% Normal Dose: number analyzed (Participants) | 27 | 25
  100% Normal Dose | 270.46 (201.73) | 307.81 (204.27)
  150% Normal Dose: number analyzed (Participants) | 27 | 25
  150% Normal Dose | 174.38 (182.00) | 123.97 (118.82)

2. Secondary Outcome: Pharmacokinetics (PK): Under the Concentration Curve Zero Through 5 Hours (AUC 0-5h) for Prandial Insulin Lispro
Description: Abbreviation for hours times picomol per liter (pmol*h/L)
Time Frame: Day 29: Pre-breakfast, and 15, 30, 45, 60, 90, 120, 150,180,210,270, and 300 minutes (5 hours) post-breakfast
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*h/L
Arm/Group | Insulin Peglispro (LY2605541) | Insulin Glargine
Number analyzed (Participants) | 23 | 21
pmol*h/L | 850 (47) | 852 (44)

3. Secondary Outcome: Pharmacodynamics (PD): Average Glucose Infusion Rate From Euglycemic 2-step Hyperinsulinemic Clamp (M-value)
Description: Abbreviation for micro mole per kilogram per minute (µmol/kg/min). Both arms received insulin lispro in addition to their respective study drug. During the euglycemic 2-step hyperinsulinemic clamp, both low and high insulin was infused sequentially during the same procedure. The 2-step clamp procedure allowed insulin sensitivity to be measured in participants and uses a lower dose of insulin of which the effect is largely on the liver and a high dose of insulin at which the effect has reached 100% on liver and effects are largely on glucose uptake in peripheral tissues. Measurements for average glucose infusion rate are collected for both steps (low and high) of the clamp procedure.
Time Frame: Day 35, last 60 minutes of euglycemic 2-step hyperinsulinemic clamp
Population: All participants who received at least 1 dose of study drug and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: µmol/kg/min
Arm/Group | Insulin Peglispro (LY2605541, With Insulin Lispro) | Insulin Glargine (With Insulin Lispro)
Number analyzed (Participants) | 12 | 11
µmol/kg/min
  High Dose Insulin | 52.756 (11.862) | 56.321 (10.697)
  Low Dose Insulin | 13.908 (13.181) | 18.765 (8.293)

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve From Time Zero to Last Time (AUC [0 Tlast]) for Paracetamol
Time Frame: Day 29: Pre-breakfast, and 15, 30, 45, 60, 90, 120, 150,180,210,270, and 300 minutes (5 hours) post-breakfast
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Insulin Peglispro (LY2605541, With Insulin Lispro) | Insulin Glargine (With Insulin Lispro)
Number analyzed (Participants) | 27 | 24
ng*hr/mL | 33400 (19) | 33600 (22)

5. Secondary Outcome: Appetite and Satiety Ratings, as Measured Using Visual Analog Scale (VAS) on Day 29
Description: VAS was scored from 0 - 100 millimeters (mm) as a perception of appetite and satiety (Flint et al. 2000), 0 being not hungry at all or nothing at all and 100 being extremely hungry and extremely large amount.
  The questions are abbreviated in table from: How hungry do you feel right now? to Hunger and How much food do you think you could eat right now? to Food amount.
  Day 29 and cumulative insulin lispro doses of 25%, 50%, 75%, 100% and 150 % of normal insulin lispro dose included.Scores were averaged will be presented and calculated by a sum of the scores dividing by the total by the number of scores reported for timepoints and reported in millimeters.
Time Frame: Day 29:Upon waking, pre-breakfast, 1 hour (hr), 2 hr, 3 hr, 4 hr and 5 hr post breakfast
Population: All participants who received at least 1 dose of study drug and had VAS score.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Groups:
- Insulin Peglispro (LY2605541, With Insulin Lispro): Insulin peglispro (LY2605541, once daily subcutaneous (SC) injection at bedtime. Insulin lispro given SC prandially or as bolus as required
Arm/Group | Insulin Peglispro (LY2605541, With Insulin Lispro) | Insulin Glargine (With Insulin Lispro)
Number analyzed (Participants) | 27 | 27
millimeters (mm)
  Day 29: Hunger, waking | 27.1 (22.1) | 32.1 (26.5)
  Day 29: Hunger, 5 hours post breakfast | 53.8 (27.9) | 58.9 (24.6)
  Day 29: Food amount, waking | 32.5 (20.6) | 37.7 (22.8)
  Day 29: Food amount, 5 hours post-breakfast | 31.8 (20.1) | 38.1 (21.8)
  Overall 25%: Hunger, waking | 27.5 (30.4) | 35.8 (28.5)
  Overall 25%: Hunger, 5 hours post breakfast | 56.1 (30.7) | 58.0 (26.2)
  Overall 25%: Food amount, waking | 30.8 (28.9) | 36.4 (27.6)
  Overall 25%: Food amount, 5 hours post-breakfast | 56.5 (28.0) | 59.0 (24.9)
  Overall 50%: Hunger, waking | 36.0 (26.2) | 28.2 (21.9)
  Overall 50%: Hunger, 5 hours post breakfast | 56.5 (26.7) | 64.0 (25.0)
  Overall 50%: Food amount, waking | 37.1 (25.2) | 31.7 (21.9)
  Overall 50%: Food amount, 5 hours post-breakfast | 55.0 (24.8) | 64.2 (23.5)
  Overall 75%: Hunger, waking | 29.8 (25.4) | 30.9 (27.5)
  Overall 75%: Hunger, 5 hours post breakfast | 55.5 (27.7) | 62.5 (25.3)
  Overall 75%: Food amount, waking | 32.6 (24.6) | 31.4 (55.3)
  Overall 75%: Food amount, 5 hours post-breakfast | 57.0 (27.1) | 62.2 (24.0)
  Overall 100%: Hunger, waking | 28.9 (22.9) | 29.6 (24.3)
  Overall 100%: Hunger, 5 hours post breakfast | 55.0 (30.2) | 59.0 (26.9)
  Overall 100%: Food amount, waking | 32.3 (22.9) | 35.7 (23.7)
  Overall 100%: Food amount, 5 hours post-breakfast | 55.3 (29.1) | 58.6 (26.4)
  Overall 150%: Hunger, waking | 31.4 (20.4) | 28.5 (16.9)
  Overall 150%: Hunger, 5 hours post breakfast | 52.2 (27.7) | 58.6 (28.4)
  Overall 150%: Food amount, waking | 34.3 (17.6) | 34.1 (17.1)
  Overall 150%: Food amount, 5 hours post-breakfast | 52.7 (25.9) | 58.3 (26.1)

6. Secondary Outcome: Pharmacodynamics (PD): Area Under the Concentration Zero Through 5 Hours (AUC 0-5h) for Triglycerides
Time Frame: Day 29, predose and 15, 30, 45, 60, 90, 120, 150,180,210,270, and 300 minutes (5 hours) post-breakfast
Population: All participants who received at least 1 dose of study drug and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Insulin Peglispro (LY2605541), With Insulin Lispro): Insulin peglispro (LY2605541) once daily subcutaneous (SC) injection at bedtime. Insulin lispro given SC prandially or as bolus as required
Arm/Group | Insulin Peglispro (LY2605541), With Insulin Lispro) | Insulin Glargine (With Insulin Lispro)
Number analyzed (Participants) | 27 | 27
ng*hr/mL | 6.85 (3.13) | 6.01 (2.22)

7. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve (AUC) for Insulin Lispro During Clamp
Description: During the euglycemic 2-step hyperinsulinemic clamp, both low and high insulin was infused sequentially during the same procedure. The 2-step clamp procedure allowed insulin sensitivity to be measured in participants and uses a lower dose of insulin (Low) of which the effect is largely on the liver and a high dose of insulin (high) at which the effect has reached 100% on liver and effects are largely on glucose uptake in peripheral tissues. AUC is taking during infusion for this outcome measure.
Time Frame: Day 35, insulin clearance during lispro infusion (dosing=infusion)
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: pmol* hr/L
Arm/Group | Insulin Peglispro (LY2605541, With Insulin Lispro) | Insulin Glargine (With Insulin Lispro)
Number analyzed (Participants) | 27 | 25
pmol* hr/L
  Clamp Period 1-3 Hours | 243 (78.9) | 222 (84.7)
  Clamp Period 4-6 Hours | 926 (335) | 897 (333)

ADVERSE EVENTS:
Description: All randomized participants.
Arm/Group | Insulin Peglispro (LY2605541, With Insulin Lispro) | Insulin Glargine (With Insulin Lispro)
Serious Adverse Events (participants affected / at risk) | 0/27 | 2/28
Other Adverse Events (participants affected / at risk) | 7/27 | 7/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Peglispro (LY2605541, With Insulin Lispro) (N=27) | Insulin Glargine (With Insulin Lispro) (N=28)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Neuralgic amyotrophy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Peglispro (LY2605541, With Insulin Lispro) (N=27) | Insulin Glargine (With Insulin Lispro) (N=28)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (7) | 4 (4)
Phlebitis (Vascular disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days